CLINICAL TRIAL: NCT03288285
Title: Effects of Post- and Pre-dilutional Hemodiafiltration on Patients With End-stage Renal Disease
Brief Title: Comparison of Post- and Pre-dilutional Hemodiafiltration in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 106042
Record Dates: First submitted 2017-09-15; First posted 2017-09-20 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Hemodiafiltration
Keywords: hemodiafiltration; pre-dilution; post-dilution; uremic toxins

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemodiafiltration (HDF) is a choice of treatment modalities for patients with end-stage renal disease. Hemodiafiltration, combining diffusion and convection, may increase removal of large and middle molecule uremic toxins comparing to conventional hemodialysis. The techniques of hemodiafiltration include pre-dilution and post-dilution according to the infusion site of substitution fluid. Post-dilution HDF is most widely used because of higher removal rate of uremic toxins. However, hemoconcentration and clotting of membrane limit its further clearance of toxins. Pre-dilution may preserve membrane permeability and maintain hemodynamic status. Although lower clearance of small molecule uremic toxins, one study in Japan showed survival benefits of pre-dilution HDF, comparing to post-dilution HDF. The aim of this study was to compare pre-dilution and post-dilution HDF in terms of their clinical and biological parameters and clearance of uremic toxins by using cross-over study design.

DETAILED DESCRIPTION:
1. Study design: randomly assigned, cross-over study.
2. Patient number: 60.
3. Inclusion criteria: stable patients end-stage renal disease who were older than 20 years and received thrice-weekly standard hemodialysis for more than 3 months were recruited.
4. Exclusion criteria: active systemic disease, liver cirrhosis, active malignancy, receiving immunosuppressive treatment, dialysis with temporal non-tunneled catheter, inadequate dialysis dose (single-pooled Kt/V<1.2).
5. Methods:

   Prior to randomization, a Charlson Comorbidity Index score and baseline characteristics are recorded for each patient. Each patient who received HDF prior to study will received one-month high-flux hemodialysis with target single-pooled Kt/V>1.2 for washout. The baseline characteristics of each patient including dialyzer, dialysis time, blood flow, dialysate flow, replacement volume, pre- and post-dialysis blood pressure and body weight were recorded. The follow-up laboratory data will also be collected: predialysis C-reactive protein, blood urea nitrogen, creatinine, bicarbonate, sodium, potassium, uric acid, albumin, calcium, phosphate, intact parathyroid hormone, β2-microglobulin, prolactin, fibroblast growth factor 23, α1-microglobulin, indoxyl sulfate, p-cresol sulfate, advance oxidation protein products, advance glycation product, percentage of proinflammatory monocytes; interleukin-6, tumor necrosis factor-α, hematocrit, transferrin saturation and ferritin. Urea kinetics including kt/V, Urea reduction ratio and normalized protein catabolic rate are calculated. We also used Physical Symptoms Distress Scale for life quality measurement.

   After randomization, two group received standard prescription of pre- and post-dilution HDF. The prescribed convective volume per treatment of post-dilution mode is based on blood flow, filtration fraction and hematocrit to achieved current recommendation of 23 liter/1.73m2. The convective volume of pre-dilution mode will be at least twice higher than the desired dose in post-dilution mode for each patient. After 3-month stable hemodiafiltration, parameters mentioned above will also be checked. Two group will be switched for another 3-month course and then switch again. The total following time is 12 months.
6. Outcome: The primary objective is to compare the removal of a wide spectrum of solutes such as middle and protein-bound molecules. Secondary outcomes are intradialytic tolerance, including intradialytic hypotension, cramps and arrhythmia, and life quality measurements.

ELIGIBILITY:
Inclusion Criteria:

* stable patients end-stage renal disease who were older than 20 years and received thrice-weekly standard hemodialysis for more than 3 months were recruited.

Exclusion Criteria:

* active systemic disease, liver cirrhosis, malignancy, receiving immunosuppressive treatment, dialysis with temporal non-tunneled catheter, inadequate dialysis dose (kt/V<1.2).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis (HD) patients
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-04-07 (Actual)

PRIMARY OUTCOMES:
Removal of a wide spectrum of solutes | 1 years
  The primary objective is to compare the removal of a wide spectrum of solutes such as middle and protein-bound molecules

SECONDARY OUTCOMES:
Intradialytic tolerance | 1 years
  intradialytic tolerance including symptomatic hypotension, cramps, headache, nutrition, and inflammatory status.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hsu Chen, MD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung Metroharbour Hospital, Taichung, Taiwan